CLINICAL TRIAL: NCT04093180
Title: Effects of Intensive Neurophysiological Rehabilitation System in Children With Cerebral Palsy: Randomized Controlled Trial
Brief Title: Intensive Neurorehabilitation for Cerebral Palsy
Acronym: IntReh4CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Clinic of Rehabilitation, Ukraine (Other)
Collaborators: I.Horbachevsky Ternopil National Medical University (Other); Elita Rehabilitation Center (Industry); Rainbow Kids e.V. (Unknown)
Responsible Party: Principal Investigator, Oleh Kachmar, Head of Innovative Techologies department, International Clinic of Rehabilitation, Ukraine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-08-03
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: Rehabilitation; Motor skills; Activities of Daily living
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group undergoing treatment course according to INRS
  Interventions: Procedure: Intensive Neurophysiological Rehabilitation System
- Control group (Other): Wait-list delayed intervention. Control group continues usual activity and care while staying in the waiting list.
  Interventions: Procedure: Activity and care as usual

INTERVENTIONS:
Procedure: Intensive Neurophysiological Rehabilitation System — Intensive Neurophysiological Rehabilitation System (INRS) is a multicomponent approach that consists of different treatment modalities.
  Arms: Experimental group
Procedure: Activity and care as usual — Control group continues usual activity and care while staying in the waiting list.
  Arms: Control group

SUMMARY:
Evaluation of effects of Intensive Neurophysiological Rehabilitation System in children with cerebral palsy in a single-blinded randomized controlled trial with two groups.

DETAILED DESCRIPTION:
Intensive Neurophysiologic Rehabilitation System (INRS) is an intensive multimodal rehabilitation system, whereby versatile and multi-faceted methods are combined with the aim of improvement of functioning and quality of life of children with CP. Treatment components are addressing different functional goals in the Body Functions domain of the International Classification of Functioning (joint mobility, muscle tone, voluntary movement, pain, intellectual functions) and Activities and Participation domains (fine hand use, walking, moving around, interpersonal interactions and family relationships.

The Intensive correction course includes up to four hours of daily training. The treatment program is tailored individually according to the patient's condition and incorporates some of the following component according to individual indications and contraindications: Physical therapy, Occupational therapy, Full body massage, Spinal manipulative therapy, Joint mobilization techniques, Paraffin and wax applications, Reflexotherapy, Strength training, Computer game therapy, Suit therapy, Vibration therapy, Treadmill training, Group session of "rhythmic gymnastics". The influence of one technique complements and potentiates other rehabilitation components.

The aim of the study is to evaluate effects of Intensive Neurophysiological Rehabilitation System in children with cerebral palsy in a randomized controlled trial.

A single-blinded randomized controlled trial with two groups will be conducted. The experimental group will undergo treatment course according to INRS, control group will continue receive usual home activity and care while staying on the waiting list. To avoid possible information leak about patient group allocation, the study should be performed in two independent centers: Evaluation center and Treatment center. Assessments will be conducted three times: at the baseline, in 3 weeks, and 7 weeks after the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy bilateral spastic forms,
* Age 4-12 years,
* Gross Motor Function Classification System - Levels I-IV,
* Manual Ability Classification System - Levels I-IV.

Exclusion Criteria:

* Uncontrolled epileptic syndrome,
* Severe intellectual disability,
* Uncooperative behavior,
* Surgery during ongoing year.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure score (GMFM-66) | Baseline, 3-week, and 7-week follow-up
  The Gross Motor Function Measure (GMFM) evaluates gross motor function in children with cerebral palsy. The GMFM-66 version contains 66 items that span the spectrum from activities as lying and rolling up to walking, running, and jumping skills.

SECONDARY OUTCOMES:
Change in Manual dexterity | Baseline, 3-week, and 7-week follow-up
  Manual dexterity is evaluated using Box and Blocks test. The score is the number of blocks carried by hand from one to another compartment in one minute.
Change in Daily functioning- Self-Care | Baseline, 3-week, and 7-week follow-up
  Eating, grooming, dressing, bathing, and toileting skills are evaluated using Pediatric Evaluation of Disability Inventory (PEDI) Self-care questionnaire that includes 73 items, scales score is calculated.
Change in Daily functioning- Mobility | Baseline, 3-week, and 7-week follow-up
  Transfers, indoor, and outdoor mobility skills are evaluated with Pediatric Evaluation of Disability Inventory (PEDI) mobility questionnaire that includes 59 items, scales score is calculated.
Change in Jebsen-Taylor hand function score | Baseline, 3-week, and 7-week follow-up
  Test quantifies the time it takes for the subject to do the following standardized functional tasks with one hand: turning over cards, picking up small items, simulating feeding, stacking checkers, picking up light cans, and picking up heavy cans.
Change in ABILHAND-Kids score | Baseline, 3-week, and 7-week follow-up
  The scale measures a person's ability to manage daily activities that require the use of the upper limbs. The parent is asked to fill in the questionnaire by estimating their child's performance of 21 manual activities on a 3-level scale (impossible, difficult, easy).
Change in passive range of ankle dorsiflexion | Baseline, 3-week, and 7-week follow-up
  Range of motion is measured with a hand-held goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Oleh Kachmar, MD, PhD, Principal Investigator — International Clinic of Rehabilitation, Ukraine
Locations (1):
- International Clinic of Rehabilitation, Truskavets, Lviv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kachmar, O. O., Mysula, I. R., Kushnir, A. D., Fedchyshyn, B. Y., & Melekh, N. V. Effect of Professor Kozyavkin method on hand function in children with cerebral palsy. International Neurological Journal. 2020;16(1): 2-9 https://doi.org/10.22141/2224-0713.16.1.2020.197324
- [Background] Kachmar, O., Mysula, I., Kushnir, A., Voloshyn, T., Matiushenko, O., Hasiuk, M., & Hordiyevych, M. (2019). Changes in motor functions in children with cerebral palsy after the course of intensive neurophysiological rehabilitation: a single-blind study. International Neurological Journal. 2019; (5): 5-11. https://doi.org/10.22141/2224-0713.5.107.2019.176700
- [Derived] Kushnir A, Kachmar O. Intensive Neurophysiological Rehabilitation System for children with cerebral palsy: a quasi-randomized controlled trial. BMC Neurol. 2023 Apr 20;23(1):157. doi: 10.1186/s12883-023-03216-4. PMID 37081406